CLINICAL TRIAL: NCT05245734
Title: Open-label, Multicenter, International Study of the Efficacy and Safety of the Drug Rhesoglobin (Human Anti-D (rh) Immunoglobulin) Manufactured by Biopharma Plasma LLC, Ukraine, in Pregnant Women in the Antenatal and Postnatal Period in Routine Clinical Practice for the Prevention of Rh Sensitization, With a Subgroup for Evaluation of Some Pharmacokinetic Parameters
Brief Title: Human Anti-D (rh) Immunoglobulin (Rhesoglobin) Efficacy, Safety and Some Pharmacokinetics Parameters in Pregnant Women
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Biopharma Plasma LLC (Industry)
Collaborators: State Institution, Zaporizhzhia Medical Academy of Post-Graduate Education Ministry of Health of Ukraine (Other); Ivano-Frankivsk National Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1901-RH-BF
Record Dates: First submitted 2022-01-06; First posted 2022-02-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related
Keywords: Rh-immunization prevention; human anti-D (rh) immunoglobulin; Rh-negative women; prenatal prophylaxis; postnatal prophylaxis
MeSH Terms: interventions — Rh-Hr Blood-Group System; Immunoglobulins

STUDY DESIGN:
Intervention Model Description: uncontrolled, open-label, multicenter, international (From the total number of patients a subgroup for studying some pharmacokinetics parameters is formed )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main group (Experimental): Patients receive two prophylactic doses of the Human Anti-D (rh) immunoglobulin at a dose of 300 mcg - at 28 weeks of gestation and within 72 hours after delivery. Patients receive the second dose only in the case of the birth of an Rh-positive child.
  Before and after each injection of the drug, blood will be taken to control the level of anti-Rh0 (D) antibodies. after the last injection of the drug, blood samples are taken after 3 and 6 months to assess sensitization to the Rh antigen.
  15 participants from the Main group are formed the "Pharmacokinetics" subgroup for additional blood samples taking, to determine the pharmacokinetic parameters
  Interventions: Drug: Human Anti-D (rh) immunoglobulin

INTERVENTIONS:
Drug: Human Anti-D (rh) immunoglobulin — prevention of Rh-sensitization in pregnant women in the antenatal and postnatal period in routine clinical practice. The study drug is administered twice at a dose of 300 mcg - at 28 weeks of gestation and within 72 hours after delivery.
  Other Names: Rhesoglobin

SUMMARY:
Rhesus conflict between mother and fetus is due to the different antigenic composition of erythrocytes. During the first pregnancy, sensitization of the mother to fetal erythrocytes rhesus D (RhD) antigens is formed. During the next pregnancy, fetal red blood cells are attacked by the mother's antibodies, and fetal/newborn hemolytic disease develops. The drug Rhesoglobin blocks the interaction of the fetal erythrocytes RhD antigen and the immune system of the mother and prevents the development of Rhesus sensitization.

DETAILED DESCRIPTION:
The screening stage The pregnant woman (participant) has to sign an informed consent. After the signed informed consent procedure, the patient is assessed for meeting the inclusion and non-inclusion (exclusion) criteria. Patients who were included in the study are assessed according to additional criteria for inclusion in the "Pharmacokinetics" subgroup.

The clinical stage

According to the study protocol, patients receive two prophylactic doses of the study drug at a dose of 300 mcg - at 28 weeks of gestation and within 72 hours after delivery. Patients receive the second dose only in the case of the birth of an Rh-positive child. Before and after each injection of the drug, blood will be taken to control the level of anti-Rh0 (D) antibodies. In the "Pharmacokinetics" subgroup, additional blood samples will be taken to determine the following pharmacokinetic parameters:

* Serum clearance
* Volume of distribution
* AUC (area under curve)
* Т1/2 (α and β) (half-life time)
* Cmax (maximum/peak serum concentration)
* Tmax (time to reach the maximum serum concentration)
* Kel (elimination rate constant)

The final stage The patient should be monitored for 6 months ± 5 days, after the last injection of the drug, blood samples are taken after 3 and 6 months to assess sensitization to the Rh antigen.

ELIGIBILITY:
Inclusion Criteria:

* Rh-negative women who are not sensitized to Rh0 (D) antigen between the ages of 18 and 45;
* signed informed patient consent to participate in the study;
* pregnancy from a Rh-positive man;
* immunocompetent patients (CD 4+ counts above 200 per μl, HIV negative, or those with the virus particle count of less than 200 per μl or 400000 per ml);
* body mass index should be within normal limits (> 18.5 kg / m2 and <30.0 kg / m2);
* patients who have not received blood transfusions and / or medicinal products containing immunoglobulins in the last 6 months, in particular antibodies to Rh0 (D) antigen;
* persons who do not have acute and chronic cardiovascular, neuroendocrine, kidney, liver diseases, diseases of gastrointestinal tract, respiratory system;
* the results of physical, instrumental and laboratory examination of patients should be within the norma or deviations should be regarded by the researcher as clinically insignificant;
* the ability, according to the researcher, to comply with all the requirements of the study protocol.

Exclusion Criteria:

* sensitization to Rh0 (D) antigen;
* the absence of reliable anamnestic data on the prevention of Rh incompatibility in previous pregnancy (s) with the birth of a Rh-positive child;
* selective IgA deficiency in the presence of antibodies against immunoglobulin A (IgA);
* history of severe allergic reactions to the administration of human blood protein preparations;
* hypersensitivity reactions to human donor immunoglobulins;
* severe thrombocytopenia and other hemostatic disorders;
* life-threatening conditions and / or complications that require intensive care / surgery, the presence of any other bleeding at the time of screening;
* Rh-negative fetus;
* any other concomitant decompensated diseases or acute conditions, the presence of which, according to the researcher, can significantly affect the study results;
* participation in any other clinical trial in the last 3 months and throughout the study.

Additional exclusion criteria:

Subgroup "Pharmacokinetics" (patients included in the additional study of some pharmacokinetic parameters):

* any previous disease or intervention that, according to the researcher, may affect the pharmacokinetics of the study drug, in particular, organ and bone marrow transplantation, cancers;
* presence of HIV, hepatitis B, or C viruses;
* presence of severe clinical and laboratory manifestations of impaired liver and kidney function

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study will include pregnant women
Enrollment: 281 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The part of patients with no antibodies to Rh0 (D) antigen | 6 months after the last administration of the drug
  The proportion of patients with no antibodies to Rh0 (D) antigen 6 months after the last administration of the drug

SECONDARY OUTCOMES:
Titer of anti-Rh0 (D) antibodies | 3 months after delivery
  Titer of anti-Rh0 (D) antibodies 3 months after delivery
Titer of anti-Rh0 (D) antibodies | 6 months after delivery
  Titer of anti-Rh0 (D) antibodies 6 months after delivery
The part of patients with no antibodies to Rh0 (D) antigen 3 months after delivery | 3 months after the last administration of the drug
  Proportion of patients with no antibodies to Rh0 (D) antigen 3 months after the last administration of the drug
Proportion of patients who developed adverse events and reactions (AE / AR) | 9 months from the first administration of the drug
  Proportion of patients who developed adverse events and reactions (AE / AR) associated with the administration of the drug, stratified by severity

OTHER OUTCOMES:
Serum clearance | 3 months after first administration of the study drug
  Pharmacokinetic parameter are determined after first administration of the study drug
volume of distribution | 3 months after first administration of the study drug
  Pharmacokinetic parameter are determined after first administration of the study drug
Area under the curve (AUC) | 3 months after first administration of the study drug
  Pharmacokinetic parameter are determined after first administration of the study drug
Half-life time (T1/2 α and β) | 3 months after first administration of the study drug
  Pharmacokinetic parameter are determined after first administration of the study drug
Maximum/peak serum concentration (Cmax) | 3 months after first administration of the study drug
  Pharmacokinetic parameter are determined after first administration of the study drug
Time to reach the maximum serum concentration (Tmax) | 3 months after first administration of the study drug
  Pharmacokinetic parameter are determined after first administration of the study drug
Elimination rate constant (Kel) | 3 months after first administration of the study drug
  Pharmacokinetic parameter are determined after first administration of the study drug

CONTACTS AND LOCATIONS:
Locations (16):
- Ukraine (16):
  - Municipal non-profit enterprise "Cherkasy Regional Hospital of Cherkasy Regional Council", Cherkasy, Cherkasy Oblast
  - Municipal non-profit enterprise "Maternity hospital" of the Chernihiv city council, Chernihiv
  - Municipal non-profit enterprise "Chernivtsi Regional Perinatal Center", Chernivtsi
  - Municipal enterprise "Dnipropetrovsk Regional Perinatal Center (DRPC) with a hospital" of the Dnipropetrovsk Regional Council, Dnipro
  - Municipal non-profit enterprise "Ivano-Frankivsk Regional Perinatal Center Ivano-Frankivsk Regional Council", Ivano-Frankivsk
  - Municipal non-profit enterprise "Khmelnytsky Regional Hospital" of the Khmelnytsky Regional Council, Khmelnytskyi
  - Municipal non-profit enterprise "Kirovohrad Regional Hospital of the Kirovohrad Regional Council", Kropyvnytskyi
  - State Institution "Institute of Pediatrics, Obstetrics and Gynecology named after academician O.M. Lukyanova National Academy of Medical Sciences of Ukraine ", Kyiv
  - Kyiv City Center for Reproductive and Perinatal Medicine, Kyiv
  - Municipal enterprise "Volyn Regional Territorial Medical Association for the Protection of Motherhood and Childhood" Volyn Regional Council, Lutsk
  - Municipal non-profit enterprise Lviv Regional Council "Lviv Regional Clinical Perinatal Center", Lviv
  - Municipal non-profit enterprise "Mykolayiv regional clinical hospital" of the Mykolayiv regional council, Mykolayiv
  - Municipal enterprise "Poltava Regional Clinical Hospital named after M.V. Sklifosovsky Poltava regional council", Poltava
  - Municipal Institution "Regional Perinatal Center" of Rivne Regional Council, Rivne
  - Municipal non-profit enterprise Sumy regional council "Regional Clinical Perinatal Center", Sumy
  - Municipal non-profit enterprise "Maternity hospital №3" of Zaporizhia City Council, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
The results will be published after trial completion. Access to parts of Clinical Study Report (CSR) planned after the release of scientific publications.
  Individual participant data (IPD) with the code of each patient will be available In CSR
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the scientific publication of trial results, 3 months later
Access Criteria: For specialists in field medicine, pharmacy, scientists

REFERENCES:
- See also: European Medicines Agency Guideline for Clinical investigation of human anti-D immunoglobulin for intravenous and/or intramuscular use, CPMP/BPWG/575/99 Rev. 1 — https://www.ema.europa.eu/en/clinical-investigation-human-anti-d-immunoglobulin-intravenous-andor-intramuscular-use